CLINICAL TRIAL: NCT02835521
Title: Influence of Perception of Patients Suffering of Osteoarthritis of Knee Over the Effectiveness and Tolerance in Intra-articular Injection of Corticoids: a Prospective, Controlled and Randomized Study
Brief Title: Influence of Perception of Patients Suffering of Knee Osteoarthritis Regarding Effectiveness of Intra-articular Injection
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Sandra Regina Toffolo, Principal Investigator, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEP UNIFESP - 849746
Record Dates: First submitted 2016-07-11; First posted 2016-07-18 (Estimated); Last update posted 2016-07-18 (Estimated); Status verified 2016-07

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Injections, Intra-Articular; triamcinolone hexacetonide

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Group (Experimental): Patients will receive the reception treatment before the joint injection
  Interventions: Procedure: Reception; Drug: Joint injection with triamcinolone hexacetonide
- Control Group (Active Comparator): patient will receive a joint injection
  Interventions: Drug: Joint injection with triamcinolone hexacetonide

INTERVENTIONS:
Procedure: Reception
  Arms: Intervention Group
Drug: Joint injection with triamcinolone hexacetonide — joint injection with corticosteroids

SUMMARY:
Introduction; reception must be understood as the offered attention within the relationship between a healthcare worker and the patient, including attitudes of inclusion, hearing, valorization of complains and identification of needs, being these individual collective. As a part of this process, communication is a primary and indispensable toll through which the healthcare team and the patient interchange information.

Objective: to evaluate the influence of perception of patients suffering of knee osteoarthritis over fear, catastrophizing of pain and effectiveness, related to intra-articular injection od corticosteroids.

Material and method: it will be performed a prospective, controlled and randomized study eith a blind evaluator on patients with symptomatic knee osteoarthritis submitted to joint injection. A hundred patients suffering of symptomatic knee osteoarthritis coming from the outpatient area of Rheumatology Division of Federal University of Sao Paulo (UNIFESP) will be evaluated, 50 belonging to the intervention group (reception) and 50 to a control group.

ELIGIBILITY:
Inclusion Criteria:

* knee osteoarthritis according to american college of rheumatology criteria
* no previous experience of joint injection
* stable use of drugs for osteoarthritis treatment for at least 3 months
* stable dose of corticosteroids, non hormonal anti-inflammatory and analgesics in the previous month
* pain on knee between 3 and 7 in the visual analogue scale
* signe the informed consent term
* radiologic classification between 1-3 (kellgren and Lawrence classification)

Exclusion Criteria:

* joint disease of different etiology
* coagulation alteration
* non treated fibromyalgia
* litigation
* diabetes mellitus and systemic arterial hypertension out of control
* allergy of lidocaine or triamcinolone hexacetonide

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-02 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Change on pain | baseline, after 1, 4 and 12 weeks
  Pain will be evaluated with an visual analogue scale

SECONDARY OUTCOMES:
Change on functional capacity | baseline, after 1, 4 and 12 weeks
  functional capacity will be evaluated with Health assesment questionary (HAQ)
Change on Catastrophizing | baseline, after 1, 4 and 12 weeks
  Catastrophizing will be evaluated with an Catastrophizing test
Change on functional capacity | baseline, after 1, 4 and 12 weeks
  functional capacity will be evaluated with the time to up and go test

IPD SHARING:
Plan to Share IPD: No